CLINICAL TRIAL: NCT05082831
Title: A Prospective, Multicenter, Randomized, Controlled Trial to Evaluate the Safety and Efficacy of a Human Extracellular Matrix Implanted in the Bone Interstices & the Cartilage Defect Following Arthroscopic Microfracture Surgery in the Knee,in Comparison to Microfracture Surgery Alone
Brief Title: Human ECM Implanted Within Microfracture Interstices & the Cartilage Defect in the Knee to Regenerate Hyaline Cartilage
Acronym: hECM;HST003
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in enrollment
Sponsor: Histogen (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HST003-ORT-001-CR
Record Dates: First submitted 2021-06-08; First posted 2021-10-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Articular Cartilage Disorder of Knee; Cartilage Damage; Microfractures
Keywords: Hyaline Cartilage; Cartilage, Articular; Arthroscopic, Subchondral; Extracellular Matrix Proteins; Extracellular Matrix; Arthroscopic Subchondral Bone Microfracture
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: This is an Intervention Model where all patients who are identified/confirmed candidates for microfracture surgery will be enrolled to receive the microfracture surgery (standard of care). Ten (10) patients will be randomized to receive the study intervention (HST003). HST003 will be injected into the microfracture defects (interstices) and fill the remainder of the defect to the cartilage margin following surgery. The primary purpose of the study is to compare the two groups: microfracture surgery + HST003 as compared to the microfracture surgery only group.
Who Masked: Participant
Masking Description: Patients will be randomized on the treatment day (Visit 2 per Schedule of Activities below) to undergo microfracture surgery with or without HST003 injection into the interstices and defect post-microfracture procedure. Each clinical site will have a study drug dispenser who will be responsible for randomizing the patient via the IWRS and will know whether the patient will be receiving HST003 or not, maintaining the blinding until the surgeon is approaching the end of the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- microfracture surgery + HST003 (Active Comparator): This is an Intervention Model where all patients who are identified/confirmed candidates for microfracture surgery will be enrolled to receive the microfracture surgery (standard of care). Ten (10) patients will be randomized to receive the study intervention (HST003). HST003 will be injected into the microfracture defects (interstices) and fill the remainder of the defect to the cartilage margin following surgery.
  Interventions: Biological: microfracture surgery + HST003
- microfracture surgery only (No Intervention): This is an Intervention Model where all patients who are identified/confirmed candidates for microfracture surgery will be enrolled to receive the microfracture surgery (standard of care). Ten (10) patients will be randomized to receive the microfracture surgery (standard of care).

INTERVENTIONS:
Biological: microfracture surgery + HST003 — This is an Intervention Model where all patients who are identified/confirmed candidates for microfracture surgery will be enrolled to receive the microfracture surgery (standard of care). Ten (10) patients will be randomized to receive the study intervention (HST003). HST003 will be injected into the microfracture defects (interstices) and fill the remainder of the defect to the cartilage margin following surgery. The primary purpose of the study is to compare the two groups: microfracture surgery + HST003 as compared to the microfracture surgery only group.
  Arms: microfracture surgery + HST003

SUMMARY:
HST003 is a human extracellular matrix designed for injection into the subchondral bone following microfracture surgery by an injection into the interstices created by the surgical awl and filling the full defect to help restore-regenerate hyaline cartilage to a pre-injury state. In this Phase 1/2 clinical trial, we will be addressing the knee joint in conjunction with microfracture surgery.

HST003 is human extracellular matrix secreted by human dermal fibroblasts under hypoxic conditions. The various matrix proteins produce a combination structural scaffold in addition to the natural secreted glycoproteins such as lubricin, fibronectin, laminins, hyaluronic acid, and collagens - all critical components of cartilage, particularly hyaline cartilage. This Phase 1/2 study will help design additional studies to support FDA approval for the use of HST003 in focal cartilage defects in the knee resulting from recent traumatic injury.

DETAILED DESCRIPTION:
HST003 belongs to a new class of natural human matrix components geared toward cartilage regeneration. The bulk of this purified hECM is structural collagens, actin, and tubulin, but it also contains structural glycoproteins. HST003 is a physiological scaffold to support the infiltration of autologous mesenchymal stem cells to regenerate cartilage, and preferably hyaline cartilage. The safety of HST003 is supported by preclinical data, which show that hECM is nontoxic, noncytotoxic, nongenotoxic, non-irritant, non-sensitizing, and non-pyrogenic. The preclinical data summary is contained in the Investigator Brochure (IB) including biocompatibility data. A description of the manufacture, chemistry, efficacy, and preclinical safety of HST003 is also provided in the IB.

The comparator in this study will be microfracture surgery alone, the current standard of care. Microfracture treatment is a single-stage arthroscopic procedure that is minimally invasive and has limited surgical morbidity (see surgical ICF for standard microfracture).

ELIGIBILITY:
Inclusion Criteria:

- Age

1. Participant must be ≥ 18 years and ≤ to 50 years of age (18-50), at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Patients who are "healthy" as determined by medical evaluation including medical history, physical exam, laboratory tests, no thyroid conditions, and no history of cancer, etc.
3. Patients with controlled hypertension defined as systolic blood pressure less than 140mmHg and diastolic blood pressure less than 90mmHg.
4. Patients with well controlled diabetes mellitus type 2 defined as an HbA1C of less than 6.5%.
5. Patients that have hematological parameters as follows: hematocrit ≥ 28.0%, white blood cell count ≤ 14,000/mm3, platelet count ≥ 50,000/mm3, creatinine

   ≤ 2.0mg/dL and International Normalized Ration (INR) ≤ 1.6.
6. Patients that have been diagnosed with a symptomatic (knee pain, effusion, and limitation of activity due to the lesion) cartilage lesion of the medial or lateral femoral condyle and have failed to respond to more conservative pharmacologic or non-pharmacologic treatments. Acute, isolated, traumatic defects are permitted in the study.
7. A cartilage lesion on the medial or lateral femoral condyle that is Grade III or IV on the Outerbridge scale, and having size of 2 cm2 - 4 cm2 as detected by MRI or recent arthroscopy if conducted in connection with this acute knee injury.
8. Intact ligaments - including intact (i) anterior cruciate ligament (ACL), (ii) lateral collateral ligament (LCL), (iii) posterior cruciate ligament (PCL), and (iv) medial collateral ligament (MCL). No concurrent ligament surgery is permitted.
9. Near normal (within 3 degrees of center) hip to ankle coronal alignment on plain radiographs. Per Schedule of Activities, X-ray of knee will be taken at screening visit.
10. Participant who is medically able to undergo knee arthroscopy and participate in the postoperative therapy protocol, including a period (up to 4 to 6 weeks) of nonweight bearing movement.
11. If participant has had prior surgery in the index knee but is stable on exam, then the participant can be included in the study (e.g., stable ACL reconstruction, diagnostic arthroscopy, plica/scar debridement, meniscus debridement less than 50%, and chondroplasty are permitted). No prior microfracture surgery in the index knee are permitted.
12. Tibial lesions on the same side as the femoral condyle lesion being treated up to Grade I or II Outerbridge grade is permitted.
13. Participant is eligible for microfracture surgery (lesion between 2cm2 - 4 cm2, Outerbridge Grade III or IV, intact subchondral plate without bony erosion, and deemed to have a clinically significant cartilage lesion).
14. Participant is able to read/write and understand the language and content of the study material, understand the requirements for follow-up visits, able and willing to comply with requirements, and is willing to provide information at the scheduled evaluations.
15. Participant is willing to use pain medication other than non-steroidal Antiinflammatory Drugs (NSAIDS) (e.g., ibuprofen/Advil and indomethacin may speed cartilage breakdown and is therefore prohibited) for 3 months post-surgery.

    Other medications (e.g., acetaminophen or narcotic analgesics) are permitted if prescribed. Post-surgical use of aspirin for clot prevention is acceptable (DVT prophylaxis acceptable) for up to 3 weeks (per surgeons standard DVT prophylaxis).
16. Participant has a creatinine clearance of more than 45 ml/min using the Cockcroft- Gault calculation.

    -Weight
17. Body mass index (BMI) greater than or equal to 18 kg/m2 and less than or equal to 35.0 kg/m2. (If patient is lean and considered healthy, yet exceeds 35.0 kg/m2, then the investigator may enroll up to 40.0 kg/m2 on a case-by-case basis).

    -Sex
18. All genders are included.

    -Informed Consent
19. Capable of giving signed informed consent as described in Section 9.1 (Appendix 1) which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

    -Inclusion of Women and Minorities in Study
20. This study will admit patients based solely on the inclusion and exclusion criteria. All potential clinical study candidates will be assessed for participation with no consideration to their gender, ethnic background or other non-pertinent classifications other than those described in the inclusion and exclusion criteria.

Exclusion Criteria:

* Medical Conditions

  1. History of substantial (greater than or equal to 50%) meniscal repair or a meniscectomy.
  2. Body Mass Index (BMI) of ≥ 35 kg/m2 and < 18 kg/m2, at the time of screening (see inclusion criteria 17 above).
  3. Known, recent (within one month of screening) history of bacterial infection regardless of body location.
  4. Prior surgical repair of the site (femoral condyle) intended to undergo microfracture surgery. No prior microfracture of the index knee is permitted.
  5. Single Assessment Numeric Evaluation (SANE) of greater than 80.
  6. Prior surgery of the contralateral knee within the last 3 months (since opposite knee needs to be intact for the non-weightbearing period post-op).
  7. Known kidney impairment, for which contrast agents for MRI could add to risks (see inclusion 16 and exclusion 13).
  8. Has vascular disorders such as varicose veins or peripheral arterial disease or neurological disorders (e.g., neuropathy affecting the index lower limb).
  9. Known allergy to anesthetics used in the study.
  10. Presence of significantly uncontrolled hypertension defined as systolic blood pressure more than or equal to 140mmHg and diastolic blood pressure more than or equal to 90mmHg.
  11. Severely uncontrolled diabetes mellitus, defined as HbA1C of 6.5% or more.
  12. Patients with results from any of the screening blood work to include: complete blood count, Prothrombin Time (PT)/Partial Thromboplastin Time (PTT)/INR, liver function, and creatinine) that exceeds 1.5 times the upper limit of normal or below 0.5 times the lower limit of normal.
  13. Patients with significant renal or hepatic impairment, as indicated by: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) greater than (>) 3 times the upper limit of normal (ULN); total bilirubin >1.5 times ULN (except in case of Gilbert's syndrome); creatinine >1.5 times ULN; hemoglobin less than (<5.5) millimole per liter (mmol/L), white blood cell count (WBC) <2.5 * 10^9 per liter, or platelets <75 *10^9 per liter).
  14. Recent (within 1 year from screening) history of thromboembolism.
  15. Known heart failure New York Heart Association (NYHA) class III or higher.
  16. Current malignancy or treatment for malignancy within the past 5 years, with the exception of non-melanoma skin cancer, or carcinoma in situ events.
  17. History of smoking (tobacco and e-cigarettes) for the previous year. No smoking throughout the trial.
  18. Known or planned pregnancy.
  19. Known allergies to rice (the recombinant human serum albumin used in the manufacturing process is produced in rice) and history of allergy to gadolinium or other contrast reagents, severe unspecified allergies or anaphylaxis.
  20. Medical conditions associated with immune suppression or medications that represent immune suppressants.
  21. Likely to need or who are currently on systemic steroids.
  22. Any other abnormal laboratory results or significant medical conditions that the Investigator believes should preclude the subject's participation in the trial.
  23. Prior surgical treatment of the index knee that remain unstable on exam, as determined by the investigator, are not permitted. Prior microfracture surgery or meniscectomy (either or both meniscus) of greater than 50% are excluded.
  24. No bone loss, no cortical disruption on MRI.
  25. Joint space narrowing of less than 3 mm on weight bearing flexion PA and standard PA radiographs. No evidence of osteophytes or significant subchondral sclerosis.
  26. History or any signs of systemic arthritis, including rheumatoid, psoriatic, ankylosing spondylitis, or other inflammatory conditions.
  27. History of or current evidence of alcohol or illicit drug dependence.
  28. Evidence on MRI of PVNS (pigmented villonodular synovitis), neoplasm, or other synovial disease.
  29. Patients unable to undergo an MRI with contrast agents or standing radiographs.
  30. History of autoimmune disease, allergic or anaphylactic disorders, hepatitis, or HIV or recent COVID-19 exposure as defined by likely exposure due to proximity to COVID-19 positive individuals and/or positive diagnosis by RT-PCR.
  31. Participant receiving therapy with anti-coagulants (including aspirin prior to surgery, heparin, coumadin, rivaroxaban, dabigatran, apixaban, edoxaban, enoxaparin, or fondaparinux) or receiving anti-platelet agents such as clopidogrel (Plavix).
  32. Has received intra-articular injection of corticosteroids, viscosupplements, PRP or stem cell therapies within the last 3 months.

      Prior/Concurrent Clinical Study Experience
  33. Current enrollment in an investigational drug or device study or participation in such a study within 30 days before enrollment.

      Other Exclusions
  34. Females with a positive pregnancy test.
  35. Is an employee of the PI/TI/EI/site or study team. Or is an employee or representative of Histogen, or a relative residing with one of the above persons.
  36. Has a condition or is in a situation which, in the TI's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.
  37. Has existing comorbidities requiring medication management either continuous or intermittent that could confound the safety and efficacy of the product.
  38. Participant is currently receiving worker's compensation or disability or is in litigation for worker's compensation or disability claims.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the KOOS (Knee Injury and Osteoarthritis Outcome Score) questionnaire | Day 168 (week 24, Visit 8)
  The KOOS (Knee Injury and Osteoarthritis Outcome Score) questionnaire will be completed at Screening (only questions 5-9 of the pain sub-form) and at Day 0 (before surgery), 42, 84, 168 and 365. Change from baseline in the KOOS pain sub-score will be compared between the study and control groups to test the hypothesis that use of HST003 in arthroscopic microfracture surgery is associated with an equal or lesser pain score than control. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL). Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms). Higher scores represent higher/better levels of function.
Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the validated IKDC (International Knee Documentation Committee) questionnaire | Day 168 (week 24, Visit 8)
  The IKDC (International Knee Documentation Committee) questionnaire will be completed at Day 0 (before surgery), 42, 84, 168, 365 and 730. Change from baseline in the IKDC score will be compared between the study and control groups to test the hypothesis that use of HST003 in arthroscopic microfracture surgery is associated with an equal or greater knee function score than control. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaire between baseline and month 6 | Day 168 (week 24, Visit 8)
  Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaire between baseline and Month 6. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Lower scores represent more pain, stiffness, and function values.
Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the Visual Analog Scale (VAS) questionnaire between baseline and month 6 | Day 168 (week 24, Visit 8)
  Assessment of joint pain equal to or lesser than microfracture alone, and equal or greater function, as measured using the Visual Analog Scale (VAS) questionnaire between baseline and Month 6. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Presence of new hyaline or fibrous cartilage formation within the repaired defects as visualized by MRI | Day 168 (week 24, Visit 8) and Day 365 (week 52, Visit 9)
  Presence of new hyaline or fibrous cartilage formation within the repaired defects as visualized by MRI at Day 168 (week 24, Visit 8) and Day 365 (week 52, Visit 9), comparing microfracture with HST003 to microfracture alone. The change in the volume of cartilage defect filling (as per MOCART) equal or more than 10 pts is a positive outcome. The cartilage filling is measured in point scale of 0-20.
Investigator assessment of functional Range of Motion (ROM) including overall strength in the knee | Day 84, Day 168, and Day 365.
  Investigator assessment of functional Range of Motion (ROM) including overall strength in the knee from baseline at Day 84, Day 168, and Day 365. Normal range of motion for Flexion is 0 to 130 degrees and for Extension is 0 to 5 degrees. Greater than 10 degrees difference would be considered good/positive outcome. Pain-free ROM, beyond what was previously captured prior to treatment and is also compared to the uninjured/untreated knee).
An independent central radiology reviewer from the Image Analysis Group (IAG) will read the MRIs, blinded. The reviewer's scores will be used in the efficacy assessment. | Day 168 (week 24, Visit 8) and Day 365 (week 52, Visit 9)
  Minimum Joint Space Width (mJSW) will be performed using IAG's Dynamika's computer aided functionality. The software will recognize the contour of the bone on X-ray and place landmarks to measure the Joint Space Width of medial and lateral joint spaces (in mm). The change in mJSW will be assessed automatically and confirmed by an experienced radiologist. Observed changes in mJSW, which are beyond the measurement error (>0.13 mm; Depuis et al. OAC 2003) will be considered positive / desirable.
An independent central radiologist from the Image Analysis Group (IAG) will blindly read the MRIs evaluate cartilage quality within the repaired defects. | Day 168 (week 24, Visit 8) and Day 365 (week 52, Visit 9)
  A radiologist will assess the cartilage quality using dGEMRIC (Delayed gadolinium enhanced MRI of cartilage). MR image will be used to draw four Regions of Interest's (ROI's) of cartilage only. The map showing changes in Gd-enhanced T1-weighted (T1Gd) will be created. The average T1 of each ROI, and of all ROI's combined will be used to compare the glycosaminoglycan content in the different knee compartments in the two groups. The lower mean T1Gd of the ROIs is desired outcome.
Participant assessment of Activities of Daily Living (ADL). | Day 168 (week 24, Visit 8) and Day 365 (week 52, Visit 9)
  Participant assessment of Activities of Daily Living (ADL). The KOOS ADL sub score is calculated as the mean score of the individual items (A1-A17) divided by 4 (the highest possible score for a single answer option) and multiplied by 100. This result is then subtracted from 100. Higher values indicate higher functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Hubka, Study Director — Histogen
Locations (5):
- United States (5):
  - Site 002, Vail, Colorado
  - Site 003, Bradenton, Florida
  - Site 001, Bethesda, Maryland
  - Site 005, State College, Pennsylvania
  - Site 004, Houston, Texas

IPD SHARING:
Plan to Share IPD: No